CLINICAL TRIAL: NCT07229534
Title: A Phase IV Clinical Trial to Evaluate the Efficacy and Safety of DA-5218 in Patients With Type 2 Diabetes Inadequately Controlled With Metformin
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DA-5218 in Patients With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA5218_DMSD_IV
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA-5218 (Experimental)
  Interventions: Drug: DA-5218
- DA-5218-C (Active Comparator)
  Interventions: Drug: DA-5218-C

INTERVENTIONS:
Drug: DA-5218 — DA-5218 + DA-5218-C placebo
  Arms: DA-5218
Drug: DA-5218-C — DA-5218-C + DA-5218 placebo
  Arms: DA-5218-C

SUMMARY:
This study is a multicenter, double-blind, active-controlled, randomized, parallel, phase IV clinical trial to evaluate the efficacy and safety of DA-5218 in patients with type 2 diabetes who have inadequate glycemic control with metformin

ELIGIBILITY:
Inclusion Criteria:

* 7.0%≤HbA1c≤10.5% and fasting glucose≤270mg/dL
* Treated with 1,000mg/day dose of metformin for at least 8 weeks

Exclusion Criteria:

* Type 1 diabetes mellitus, secondary diabetes mellitus or gestational diabetes mellitus
* eGFR<45mL/min/1.73m2
* ALT and AST 3 times or higher than upper normal range
* Determined by investigator as unfit to participate in a clinical trial due to other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of HbA1c(%) | 24 weeks